CLINICAL TRIAL: NCT02904109
Title: Randomized Placebo Controlled Phase II Cross Over Study on the Influence of Triflusal on Cognitive Functions in Subjects Under Chronic Stress
Brief Title: Influence of Triflusal on Cognitive Functions in Subjects Under Chronic Stress
Acronym: Tricross-Basel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2016DR2116
Record Dates: First submitted 2016-09-12; First posted 2016-09-16 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — triflusal; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum/Placebo (Experimental): This group will start with triflusal and after washout will receive placebo.
  Interventions: Drug: Triflusal; Drug: Placebo
- Placebo/Verum (Experimental): This group will start with placebo and will receive triflusal after washout.
  Interventions: Drug: Triflusal; Drug: Placebo

INTERVENTIONS:
Drug: Triflusal — Once daily oral administration of 600 mg triflusal Disgren® for 8 days.
  Other Names: Disgren®
Drug: Placebo — Once daily oral administration of placebo mannitol for 8 days.
  Other Names: mannitol

SUMMARY:
The purpose of this study is to investigate the effects of the eNOS activating agent triflusal on episodic memory and cognitive functions in participants under chronic stress.

DETAILED DESCRIPTION:
Randomised, placebo controlled, double blind, cross-over design

Primary study outcome is:

Performance in a verbal memory task.

Main secondary outcomes are: Performance in working memory and cognitive tasks and influence on mood, depression and anxiety and subjective memory impairment.

Once daily oral administration of 600 mg triflusal and placebo mannitol for 8 days in a cross-over trial with a washout period of at least 14 days between the two periods. Each participant will take triflusal as well as placebo

ELIGIBILITY:
Inclusion Criteria:

* male or female
* normotensive (BP between 90/60mmHg and 140/90mmHg)
* BMI between 19 and 29 kg/m2
* aged between 18 and 40 years
* experiencing chronic stress for at least 1 month (TICS sum score in subscale "overextension at work" >= 55)
* native or fluent German-speaking
* able and willing to give written informed consent as documented by signature and comply with the requirements of the study protocol
* willing to donate saliva sample for DNA-analysis
* female: willing to perform a pregnancy test at the beginning of both medication phase and at the follow-up visit.

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to salicylates and other NSAIDs
* acute or chronic psychiatric disorder (e.g. major depression, psychoses, somatoform disorder, suicidal tendency) except symptoms of chronic stress
* cognitive impairment as detected by DemTect
* concomitant acute or chronic disease state (e.g. renal failure, hepatic dysfunction, cardiovascular disease, acute infections etc.)
* women who are pregnant or breast feeding
* intention to become pregnant during the course of the study
* lack of safe contraception, defined as: female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases
* active peptic ulcer or antecedents or complicated peptic ulcer or history of peptic ulcer. Any other active pathological bleeding
* history of coagulation abnormality
* thyroid problems
* laboratory exclusion criteria: clinically significant values of blood count (incl. platelets), coagulation status or blood chemistry outside reference range of laboratory
* pathological ECG
* known or suspected non-compliance, drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* participation in another study with investigational drug within the 30 days preceding -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Change in performance in episodic memory task as assessed by a verbal memory task between placebo and verum at two different time points. Verbal task as described in ( de Quervain, Henke et al. 2003). Number of correctly * | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  Verbal task as described in ( de Quervain, Henke et al. 2003). Number of correctly remembered words is counted.

SECONDARY OUTCOMES:
Change in performance in working memory task between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  Working memory as assessed by digit span task. Number of correctly remembered digitsis counted.
Change in performance in episodic memory task between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  Episodic memory is assessed by the visual/spatial and verbal memory test VVM (Building und roadmap) (Quiske 2000). Number of correct answers is counted
Change in performance in a memory game between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  A memory game consisting of 12 pictures will be used to assess episodic memory.Total score is calculated by summing the correctly located pictures after 3 rounds of the game
Change in subjective memory impairment between placebo and verum | 20 min before last medication of each placebo and verum
  a two part questionnaire (MIQ) consisting of a 10-item Rasch modeled Memory self-efficacy scale (Zelinski and Gilewski 2004) extended by 6 items as second part.Total score is calculated by summing the answers of each part.
Mood state changes between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  Mood state as assessed by self-rating instrument MDBF. Total score is calculated by summing the answers of nine items.
Changes in depressive symptoms between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  Depressive symptoms as assessed by self-rating instrument MADRS. Total score is calculated by summing the answers of nine items.
Changes in anxiety symptoms between placebo and verum at two different time points. | Timepoint 1:45 minutes after first medication. Timepoint 1:45 minutes after last medication.
  Anxiety symptoms as assessed by self-rating instrument STAI-G from X1 (state). Total score is calculated by summing the answers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Basel, Switzerland